CLINICAL TRIAL: NCT05562557
Title: A Regional Partnership for New York City to Improve Well-Being and Child Welfare Outcomes Among Families at Risk of Substance Misuse Through Fatherhood Engagement
Brief Title: A Regional Partnership to Improve Outcomes Through Fatherhood Engagement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-14401
Record Dates: First submitted 2022-09-26; First posted 2022-09-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Substance Use; Child Abuse; Child Neglect; Fathers; Father-Child Relations
MeSH Terms: conditions — Substance-Related Disorders | interventions — Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Services as Usual (No Intervention): Randomly assigned to receive services as usual
- Enhanced Fatherhood Services through Regional Partnership Grant Round 7 (RPG7) (Experimental): Randomly assigned to receive enhanced RPG7 services (motivational enhancement, fatherhood engagement services, contingency management, case management)
  Interventions: Behavioral: Motivational Enhancement; Behavioral: HERO Dads Fatherhood Program; Behavioral: Contingency Management; Behavioral: Case Management

INTERVENTIONS:
Behavioral: Motivational Enhancement — To encourage intrinsic motivation to engage in fatherhood activities
  Arms: Enhanced Fatherhood Services through Regional Partnership Grant Round 7 (RPG7)
Behavioral: HERO Dads Fatherhood Program — Fatherhood engagement curriculum to increase awareness, knowledge, and skills for parenting and co-parenting
  Arms: Enhanced Fatherhood Services through Regional Partnership Grant Round 7 (RPG7)
Behavioral: Contingency Management — To reinforce healthy behaviors, including attendance at services
  Arms: Enhanced Fatherhood Services through Regional Partnership Grant Round 7 (RPG7)
Behavioral: Case Management — Referrals to treatment, social services, and employment services
  Arms: Enhanced Fatherhood Services through Regional Partnership Grant Round 7 (RPG7)

SUMMARY:
Montefiore will engage fathers in families at risk of substance misuse in the Bronx and neighboring communities. Families will be referred from Bronx and neighboring community-based child welfare systems, substance use disorder (SUD) treatment providers, and medical providers if identified at risk of substance use concerns and will be randomly assigned to receive services as usual as part of the comparison group, or to receive enhanced services as part of the program group.

Enhanced services include: (1) Motivational Enhancement; (2) referral to Healthy, Empowered, Resilient, and Open (HERO) Dads fatherhood engagement program; (3) Contingency Management; and (4) Case Management.

ELIGIBILITY:
Inclusion Criteria:

* (i) is a custodial or non-custodial father,
* (ii) who has at least one child under the age of 18,
* (iii) someone in the family is identified as at-risk for substance use

Exclusion Criteria:

* The placement of all children in the family in foster care

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — As this project is about fatherhood, only those who identify as fathers will be included.
Enrollment: 240 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Child well-being, as measured by: Child Behavior Checklist | Baseline
  This is a standardized self-report measure widely used in the measure of child behavior and child well-being. A separate form is used for children aged 1.5-5, and 6-18. The questionnaire is completed by the caregiver using a series of Likert scales (0=absent, 1=sometimes, 2=often occurs). There are 113 questions, measuring a series of internalizing (e.g., anxious/ depressed, depressed, somatic complaints) and externalizing (e.g., attention problems, rule-breaking behavior, aggression) symptoms over the prior 6-months. Raw scores are standardized into t-scores, with elevated scores reflecting greater symptomatology when compared to a gender and aged normed population.
Child well-being, as measured by: Child Behavior Checklist | Follow Up (6-months after Baseline)
  This is a standardized self-report measure widely used in the measure of child behavior and child well-being. A separate form is used for children aged 1.5-5, and 6-18. The questionnaire is completed by the caregiver using a series of Likert scales (0=absent, 1=sometimes, 2=often occurs). There are 113 questions, measuring a series of internalizing (e.g., anxious/ depressed, depressed, somatic complaints) and externalizing (e.g., attention problems, rule-breaking behavior, aggression) symptoms over the prior 6-months. Raw scores are standardized into t-scores, with elevated scores reflecting greater symptomatology when compared to a gender and aged normed population.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Wetzler, PhD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
No current plan. May be possible to provide individual data (de-identified) for secondary data analysis.